CLINICAL TRIAL: NCT00397904
Title: Phase II Trial of Cetuximab Plus Cisplatin and Irinotecan in Patients With Irinotecan and Cisplatin-Refractory Metastatic Esophageal and Gastric Cancer
Brief Title: Cetuximab, Cisplatin, and Irinotecan in Treating Patients With Metastatic Esophageal Cancer, Gastroesophageal Junction Cancer, or Gastric Cancer That Did Not Respond to Previous Irinotecan and Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-095; P30CA008748 (NIH); MSKCC-06095
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; recurrent esophageal cancer; recurrent gastric cancer; adenocarcinoma of the stomach; stage IV esophageal cancer; stage IV gastric cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab; Cisplatin; Irinotecan; Immunohistochemistry; Biopsy

ARMS (1):
- Cetuximab, Cisplatin, and Irinotecan (Experimental): Cetuximab will be combined with weekly irinotecan and cisplatin. Patients will receive cetuximab 400 mg/m2 on day 1, week 1. Following this loading dose, patients will receive weekly cetuximab 250 mg/m2 (day 8, 15, 22, etc.) until disease progression or unacceptable toxicity. Patients will continue to receive irinotecan and cisplatin weekly on day 1 and day 8, on an every 21 day cycle. The standard maximum doses are irinotecan 65 mg/m2 and cisplatin 30 mg/m2.
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: irinotecan hydrochloride; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: biopsy

INTERVENTIONS:
Biological: cetuximab
Drug: cisplatin
Drug: irinotecan hydrochloride
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for their growth. Drugs used in chemotherapy, such as cisplatin and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with cisplatin and irinotecan may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with cisplatin and irinotecan works in treating patients with metastatic esophageal cancer, gastroesophageal junction cancer, or gastric cancer that did not respond to previous irinotecan and cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with irinotecan hydrochloride- and cisplatin-refractory metastatic esophageal, gastroesophageal junction, or gastric cancer treated with cetuximab, cisplatin, and irinotecan hydrochloride.

Secondary

* Determine the median survival of patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.
* Determine the adverse event profiles in patients treated with this regimen.
* Assess epidermal growth factor receptor expression in tumor tissue from patients treated with this regimen.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive cetuximab IV over 60-120 minutes on days 1, 8, and 15 and cisplatin IV over 30 minutes and irinotecan hydrochloride IV over 30-90 minutes on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor biopsy at baseline to evaluate epidermal growth factor receptor by immunohistochemistry.

After completion of study treatment, patients are followed every 3 months for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Adenocarcinoma or squamous cell carcinoma of the esophagus
  * Adenocarcinoma of the gastroesophageal junction
  * Adenocarcinoma of the stomach
* Metastatic disease
* Measurable disease by diagnostic CT scan or MRI
* Failed prior treatment with cisplatin and irinotecan hydrochloride, defined by the following:

  * Radiographic progression within 12 weeks* from the last dose of prior cisplatin and irinotecan hydrochloride, administered either as adjuvant or neoadjuvant therapy, OR as therapy for metastatic disease NOTE: *Prior irinotecan hydrochloride and cisplatin must have been administered within the past 12 weeks; other chemotherapy regimens may have been administered between the time of disease progression or prior irinotecan hydrochloride/cisplatin and study entry
* Pathologic tissue available for immunohistochemistry (IHC) staining for the epidermal growth factor receptor (EGFR)

  * Positive or negative EGFR by IHC allowed

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 3 months
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin normal
* AST and ALT < 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior severe infusion reaction to a monoclonal antibody
* No history of allergic reactions to compounds of similar chemical or biologic composition to irinotecan hydrochloride, cisplatin, or other study agents
* No prior intolerance to irinotecan hydrochloride or cisplatin despite prior dose attenuations
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection requiring parenteral antibiotics
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled hypertension
  * Clinically significant cardiac arrhythmia
  * Myocardial infarction within the past 6 months
  * HIV infection
  * Psychiatric illness or social situations that would preclude study compliance
* No history of Gilbert's disease
* No medical condition or reason that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy or radiotherapy and recovered
* No more than 2 prior treatment regimens for metastatic disease
* No prior therapy specifically and directly targeting the epidermal growth factor receptor pathway
* No prior anticancer murine or chimeric monoclonal antibody therapy

  * Prior humanized monoclonal antibody therapy allowed
* No concurrent antiseizure medications known to affect the metabolism of irinotecan hydrochloride, including phenytoin or phenobarbital
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab, Cisplatin, and Irinotecan
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab, Cisplatin, and Irinotecan
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Complete and Partial Response Rate
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Cetuximab, Cisplatin, and Irinotecan
Number analyzed (Participants) | 16
participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 4
  Progression of Disease | 11

ADVERSE EVENTS:
Arm/Group | Cetuximab, Cisplatin, and Irinotecan
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab, Cisplatin, and Irinotecan (N=16)
Blood bilirubin increased (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Sudden death NOS (General disorders) | 1 (1)
Death-Disease Progression NOS (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab, Cisplatin, and Irinotecan (N=16)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (22)
Alkaline phosphatase increase (Investigations) | 3 (10)
Cardiac troponin I increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fatigue (General disorders) | 6 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (34)
INR increased (Investigations) | 2 (10)
White blood cell decreased (Investigations) | 3 (5)
Lymphocyte count decreased (Investigations) | 7 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (32)
Neutrophil count decreased (Investigations) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 (8)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes